CLINICAL TRIAL: NCT04733209
Title: Investigation of the Effectiveness of Movement With Mobilization Technique for Carpal Tunnel Syndrome.
Brief Title: Mobilization With Movement in Carpal Tunnel Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İSMAİL CEYLAN (Other)
Responsible Party: Sponsor-Investigator, İSMAİL CEYLAN, Head of hand therapy clinic. PhD., Ahi Evran University Education and Research Hospital
Organization: Ahi Evran University Education and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1206845174
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Pain, Chronic
Keywords: Pain; Mobilisation
MeSH Terms: conditions — Chronic Pain; Pain | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilization with movement (Experimental): Mobilization with movement technique and traditional physiotherapy were applied to the intervention group. For mobilization with movement technique, the patient was asked to actively flex and extend the wrist with the forearm in neutral in a sitting position on a treatment table, and the pain was asked. The painful side was determined according to the patient's statement.
  In a patient whose painful side was flexion, the wrist joint was shifted manually (with the help of the web space of both hands of the therapist) to the lateral and medial at the same time while the patient actively flexed the wrist. The treatment was done 3 times a week for 4 weeks.
  Interventions: Other: TENS, US, exercise
- Conventional (Active Comparator): Traditional physiotherapy techniques were applied to the intervention group. Conventional TENS type was used. Current transition time was set as 50-100 µs. TENS application is performed at a frequency of 100 Hertz for 20 minutes in amplitude that does not cause muscle contraction in the patient and creates a feeling of numbness and tingling. Continuous ultrasound type was applied with full contact technique. Ultrasound treatment was applied over the transverse carpal ligament in the wrist with circular movements towards the proximal and distal at a speed of 1-2.5 cm per second, at a dose of 1 W / cm2, for 6 minutes, with a frequency of 3 MHz. And; tendon-nerve gliding exercises, night splint, stretching and strengthening exercises applied. The treatment was done 3 times a week for 4 weeks.
  Interventions: Other: TENS, US, exercise

INTERVENTIONS:
Other: TENS, US, exercise — Physiotherapy

SUMMARY:
Peripheral nerve impingement neuropathies are the most common mononeuropathies encountered in clinical practice. Carpal Tunnel Syndrome (CTS) occurs as a result of compression of the median nerve as it passes through the carpal tunnel, a narrow osteofibrous canal. CTS is the most common entrapment neuropathy of the upper extremity, affecting approximately 3% of the general population.

Massage and mobilization techniques are used in the treatment of CTS due to their analgesic effects. The painless mobilization with movement technique (MWM, developed by Brian Mulligan) is a manual therapy method applies to correct the limitation of movement in the joint and to relieve pain and functional disorders. Many studies have shown that MWM technique provides faster and momentary painless joint movement compared to other physical therapy modalities.

The patient group with CTS has a large place in the general population and long treatment processes cause both labour loss and economic loss. In the literature review, there is no study examining the effects of MWM in patients with CTS. Therefore, this study aimed to examine the effectiveness of MWM technique in cases with CTS.

DETAILED DESCRIPTION:
In this study, 45 CTS patients with age range 18-65 who applied to Kırşehir Ahi Evran University Training and Research Hospital were examined. The individuals included in the study were divided into two groups according to the paired randomization method. These groups were control and intervention groups. Traditional physiotherapy methods were applied to the control group, traditional physiotherapy and MWM techniques were applied to the intervention group. Traditional physiotherapy methods were included; Transcutaneous Electrical Nerve Stimulation (TENS), Ultrasound (US), tendon-nerve gliding exercises, night splint, stretching and strengthening exercises.

For the evaluation of patients; Visual Analogue Scale (VAS), wrist goniometric measurements, grip strength measurement, pinch strength measurement, edema measurement, Electromyography (EMG), Nelson Hand Reaction Test, Upper Limb Disorders Arm Shoulder and Hand Problems Questionnaire (DASH), Boston Carpal The Tunnel Injury Questionnaire and Michigan Hand Result Questionnaire (MHRQ) was used.

ELIGIBILITY:
Inclusion Criteria:

* Lasting longer than six weeks in the area associated with the n. medianus; Paresthesia, pain, and vasomotor symptoms.

A positive Phalen, Tinel or carpal compression test on wrist examination. In neurophysiological evaluation mild to moderate severity of the n. medianus lesion

Exclusion Criteria:

* • Radial or ulnar nerve sensory-motor findings accompanying the current condition. Under the age of 18 and over the age of 65.

  * Having undergone upper extremity surgery or steroid injection for any reason. Having a history of another disease or trauma in the upper extremity.
  * Having a history of systemic disease such as diabetes or thyroid disease, which may lead to CTS.

Pregnancy.

* Any contraindications for the patient to exercise,
* The patient has any mental problems.
* In neurophysiological evaluation severe n. medianus lesion severity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-12-28 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
The disabilities of the arm, shoulder and hand (DASH) questionnaire | 0-4 week
  The disabilities of the arm, shoulder and hand (DASH) questionnaire is a self-administered region-specific outcome instrument developed as a measure of self-rated upper-extremity disability and symptoms. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100.
Visual Analogue Scale (VAS) | 0-4 week
  A Visual Analogue Scale (VAS) is a measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

SECONDARY OUTCOMES:
The Michigan Hand Outcomes Questionnaire (MHQ) | 0-4 week
  The MHQ is a patient-rated questionnaire, which means the patients evaluate their health state themselves. It was developed using the psychometric principles for psychological assessments (Reliability, Validity, Standardization, and Freedom from bias). The questionnaire consists of 37 items that can be grouped into six main categories (scored 0 (no disability) to 100). Special to this assessment is the inclusion of items about aesthetics, which is often regarded as very important by patients, and the separate evaluation of the left and the right side. These two categories are often overlooked in other similar assessments which might e.g. focus more on the overall disability or pain experience. The questions are directed towards patients' experiences with the hand/upper extremity during the past week.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Ceylan, PhD., Principal Investigator — Kirsehir Ahi Evran Universitesi
Locations (1):
- Kırşehir Ahi Evran Üniversitesi, Kırşehir, İç Anadolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beselga C, Neto F, Alburquerque-Sendin F, Hall T, Oliveira-Campelo N. Immediate effects of hip mobilization with movement in patients with hip osteoarthritis: A randomised controlled trial. Man Ther. 2016 Apr;22:80-5. doi: 10.1016/j.math.2015.10.007. Epub 2015 Oct 31. PMID 26559319
- [Result] Cruz-Diaz D, Lomas Vega R, Osuna-Perez MC, Hita-Contreras F, Martinez-Amat A. Effects of joint mobilization on chronic ankle instability: a randomized controlled trial. Disabil Rehabil. 2015;37(7):601-10. doi: 10.3109/09638288.2014.935877. Epub 2014 Jul 3. PMID 24989067
- [Derived] Ceylan I, Buyukturan O, Aykanat O, Buyukturan B, Sas S, Ceylan MF. The effectiveness of mobilization with movement on patients with mild and moderate carpal tunnel syndrome: A single-blinded, randomized controlled study. J Hand Ther. 2023 Oct-Dec;36(4):773-785. doi: 10.1016/j.jht.2023.02.004. Epub 2023 Aug 11. PMID 37573157
- See also: The official international web site — https://bmulligan.com/